CLINICAL TRIAL: NCT03947073
Title: Gestation Diabetes N'Teractive Media-based Education (GDnME) Trial
Brief Title: Gestation Diabetes N'Teractive Media-based Education (GDnME)
Acronym: GDnME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AAAR9927
Record Dates: First submitted 2019-02-25; First posted 2019-05-13 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Gestational Diabetes
Keywords: Media; Education; Gestational diabetes; Pregnancy
MeSH Terms: conditions — Diabetes, Gestational | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): Subjects with newly diagnosed gestational diabetes are randomized to standard of care diabetes education.
- Interactive Educational Application (Experimental): Subjects with newly diagnosed gestational diabetes are randomized to standard of care plus an interactive educational application.
  Interventions: Other: Education

INTERVENTIONS:
Other: Education — Three cartoon illustrated educational videos with information on gestational diabetes will be provided to the patient in addition to standard of care.
  Arms: Interactive Educational Application

SUMMARY:
This study is a prospective randomized controlled trial. Subjects with newly diagnosed gestational diabetes will be randomized to either standard of care diabetes education versus standard of care plus an interactive educational application.

DETAILED DESCRIPTION:
Gestational diabetes is a condition diagnosed during pregnancy that causes blood sugars to rise. Diet and exercise can effectively control blood sugar levels in 70-85% of women diagnosed with gestational diabetes according to the American Diabetes Association. At the investigator's institution, only 50-54% of women with this diagnosis effectively reach the target blood sugar levels with diet and exercise alone. This has become a more commonly seen problem throughout the US. Those that fail to achieve target blood sugar levels require medication and have higher risks of poor maternal and neonatal outcomes. Studies have shown that an increase in education can increase compliance to diet and education. Specifically, media based education that are interactive may more effectively lead to changes in a person's behavior.

ELIGIBILITY:
Inclusion Criteria:

* Obtaining prenatal care in the Ambulatory Care Network (ACN)
* Speaks either English or Spanish
* Newly diagnosed with gestational diabetes between 24-32 weeks
* Will deliver at CUIMC's main institutions, Children's Hospital of New York (CHONY) or the Allen Hospital.

Exclusion Criteria:

* Diagnosed with a fetal anomaly
* Have multiple gestation
* Known diagnosis of pregestational diabetes

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 199 (Actual)
Dates: Start 2019-06-12 (Actual); Primary Completion 2021-01-27 (Actual); Study Completion 2021-01-27 (Actual)

PRIMARY OUTCOMES:
Total number of women who failed management with diet alone | Up to 42 weeks
  This is defined as a patient who is unable to adequately control blood sugars with diet alone and requires medical intervention. This information will be collected until the time of delivery which could be up to 42 weeks of gestation.

SECONDARY OUTCOMES:
A1C Level | Up to 42 weeks
  A1C level will be measured at the 24-28 weeks and at approximately 37 weeks or time of delivery (up to 42 weeks).
Average fasting blood sugar level | Up to 42 weeks
  Fasting blood sugar level will be measured at first week of entry and at approximately 37 weeks or time of delivery (up to 42 weeks of gestation).
Average 2 hour post-prandial blood sugar level | Up to 42 weeks
  The 2-hour post-prandial blood sugar level (after breakfast, lunch, and dinner) will be measured at first week of entry and at approximately 37 weeks or at the time of delivery (up to 42 weeks of gestation).
Total insulin requirement | Up to 42 weeks
  Average insulin required will be measured at first week of entry and at approximately 37 weeks or at the time of delivery (up to 42 weeks of gestation).
Total metformin requirement | Up to 42 weeks
  Average metformin required will be measured at first week of entry and at delivery (up to 42 weeks of gestation).
Total number of women who develop gestational hypertension | Up to 42 weeks
  Gestational hypertension is defined as blood pressures captured after 20 weeks of gestation that are either 140 systolic or 90 diastolic on 2 occasions at least 4 hours apart. This will be collected until delivery which may be up to 42 weeks of gestation.
Total number of women who develop pre-eclampsia | Up to 42 weeks
  Pre-eclampsia is defined as blood pressures of 140 systolic or 90 diastolic on 2 occasions at least 4 hours apart during the gestation plus either neurologic/hepatic/or end organ dysfunction or proteinuria defined as protein:creatinine ratio of >0.3 or 24 hr urine protein of over 300 mg/24 hours. This will be collected until delivery which may be up to 42 weeks of gestation.
C-section rate | Up to 42 weeks
  Total number of women who have a c-section of the total number of deliveries. This will be collected until delivery which may be up to 42 weeks of gestation.
Difference in weight | Up to 42 weeks
  Weight difference from the time of diagnosis compared to weight at delivery will be measured. This will be collected until delivery which may be up to 42 weeks of gestation.
Total number of neonates with shoulder dystocia | Up to 42 weeks
  Complication during delivery when an infants shoulder's get lodged in the mother's pelvis, requiring special maneuvers in order to dislodge the shoulder. This will be collected until delivery which may be up to 42 weeks of gestation.
Total number of neonates with a NICU admission | Up to postpartum day 7
  Measures admission to the neonatal intensive care unit within 2 weeks of birth. This information will be collected until postpartum day 7.
Total number of neonates with neonatal hypoglycemia | Up to postpartum day 7
  Measures plasma glucose level of less than 30 mg/dL (1.65 mmol/L) in the first 24 hours of life and less than 45 mg/dL (2.5 mmol/L) thereafter
Total number of neonates with neonatal respiratory distress syndrome | Up to postpartum day 7
  Clinical diagnosis made by neonatologist/pediatrician: Symptoms and signs of RDS include rapid, labored, grunting respirations appearing immediately or within a few hours after delivery, with suprasternal and substernal retractions and flaring of the nasal alae. As atelectasis and respiratory failure progress, symptoms worsen, with cyanosis, lethargy, irregular breathing, and apnea. Diagnosis of RDS is by clinical presentation, including recognition of risk factors; ABGs showing hypoxemia and hypercapnia; and chest x-ray. Chest x-ray shows diffuse atelectasis classically described as having a ground-glass appearance with visible air bronchograms; appearance correlates loosely with clinical severity.
Total number of neonates with jaundice | Up to postpartum day 7
  The total number of neonates needing phototherapy to treat jaundice will be measured.
Total number of neonates with an Apgar score <7 | Up to 42 weeks
  The total number of neonates with an Apgar score of <7 at 5 minutes from birth will be measured. This information will be collected until delivery which may be up to 42 weeks of gestation.
Total number of neonates with a preterm birth | Up to 36 weeks and 6 days of gestation
  The total number of neonates with birth with a gestational period of less than 37 weeks (iatrogenic and spontaneous) will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Noelia Zork, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
yes
Supporting Information: Study Protocol, SAP
Time Frame: At the time of study completion
Access Criteria: Only information that is de-identified can be shared. Information will only be available at the end of the study period in the event that a peer review journal requests the information.